CLINICAL TRIAL: NCT00005510
Title: Strong Heart Study Analyses Obesity and Lipoproteins
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5028; R03HL060018 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2001-11

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Obesity

SUMMARY:
To examine the relationship of obesity and body fat distribution to lipoprotein concentrations in members of the Strong Heart Study.

DETAILED DESCRIPTION:
BACKGROUND:

The Strong Heart Study is a longitudinal cohort study of several American Indian groups in three participating centers. The overall aim of the main study is to determine the role of various risk factors in the development of cardiovascular disease in this native American population.

DESIGN NARRATIVE:

Data from the first and second clinical exams of the Strong Heart Study were analyzed to determine if body fat distribution as measured by waist-to-hip circumference was a better correlate of lipoproteins than was body mass index. In addition, change in body mass index (BMI) and waist-to-hip ratio (WHR) were correlated with change in lipoproteins.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-04; Study Completion 1999-03 (Actual)